CLINICAL TRIAL: NCT02095405
Title: A Prospective Placebo Controlled Randomized Study of Caffeine in Patients With Supraventricular Tachycardia Undergoing Electrophysiologic Testing.
Brief Title: A Study of Caffeine on Cardiac Arrhythmias
Acronym: CACOA-HEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Robert Lemery, Cardiac Electrophysiologist, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009403-01H
Record Dates: First submitted 2014-03-18; First posted 2014-03-24 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Supraventricular Tachycardia (SVT); Atrial Fibrillation
Keywords: Supraventricular Tachycardia; Atrial Fibrillation; Electrophysiology Study; Programmed Electrical Stimulation
MeSH Terms: conditions — Tachycardia, Supraventricular; Atrial Fibrillation | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caffeine arm (Active Comparator): SVT group: Caffeine tablets, 5 mg/kg.
  AF group: Caffeinated substances and Dark Chocolate
  Interventions: Drug: Caffeine
- Placebo arm (Placebo Comparator): SVT group: Placebo
  AF group: Decaffeinated substances and White Chocolate
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Caffeine — SVT group: Oral tablets of Caffeine prior to the electrophysiology study in patients with SVT.
  AF group: Dark chocolate and Caffeinated substances in patients with AF at the time of Ambulatory monitoring.
  Arms: Caffeine arm
Other: Placebo — SVT group: Oral tablets of placebo prior to the electrophysiology study in patients with SVT.
  AF group: White chocolate and Decaffeinated substances in patients with AF at the time of Ambulatory monitoring.
  Arms: Placebo arm

SUMMARY:
Stimulants and drugs are often associated with cardiac effects. Caffeine, a therapeutic xanthine, has been described as a sympathomimetic and has shown to have stimulatory effects on the heart. Patients with symptomatic cardiac arrhythmias are generally informed by their physician to stop or significantly reduce caffeine intake. However, in spite of numerous reports that have reviewed the cardiac effects of caffeine, it remains unclear to what extent this stimulant may be detrimental, and what subgroups of patients may be most vulnerable. The investigators propose to evaluate the effects of caffeine in patients with previously diagnosed cardiac arrhythmias. The results of our report will provide important new information for physicians and patients regarding the effects of caffeine on symptomatic cardiac arrhythmias.

DETAILED DESCRIPTION:
Caffeine is one of the most frequently consumed pharmacologic active substances in the world. The potential effects of caffeinated beverages and chocolate on human health remains of great interest. The increased prevalence of cardiac arrhythmias in the general population has resulted in greater concern about the potential effects of caffeine on cardiac arrhythmias. Patients diagnosed with a cardiac dysrhythmia are generally informed by their physician to restrict or even abstain from caffeine, despite a lack of evidence of this causal relationship.

Although there have been numerous reports published on the effects of caffeine on human health, there have been few reports on the relation between caffeinated beverages and chocolate in different subgroups of patients with previously diagnosed cardiac arrhythmias, including supraventricular tachycardia (SVT), atrial fibrillation (AF), atrial flutter, and ventricular arrhythmias. These patients frequently undergo interventional ablation procedures, and have a potential for a recurrence of their arrhythmia. A greater knowledge of the effects of caffeine in different subgroups of patients with cardiac arrhythmias is thus essential to properly guide patients and physicians in their treatment.

The objective of our study is to evaluate the effects of caffeine through noninvasive and/or invasive means on patients with documented symptomatic cardiac arrhythmias.

One group will consist of 80 patients with Supraventricular Tachycardia (SVT): This group will undergo Invasive testing, which will be completed in the electrophysiology laboratory prior to their ablation procedure to evaluate the electrophysiologic effects of caffeine or placebo on the human heart. This testing will include a measure of the effective refractory periods, inducibility of tachyarrhythmias, and conduction intervals during programmed electrical stimulation.

The other group will consist of up to 80 patients with Atrial Fibrillation: This group will undergo non-invasive testing, consisting of two consecutive 48-hr Ambulatory monitors while they consume caffeinated or noncaffeinated products.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years.
* Document cardiac arrhythmia, consisting of either:

  i. Patients with SVT: Patients with documented narrow complex tachycardia on a twelve lead ECG or on ambulatory monitoring ii. Patients with AF, paroxysmal (self-terminating AF within 7 days), documented on a twelve lead ECG or on ambulatory monitoring

Exclusion Criteria:

* Failure to provide informed consent
* Pregnancy as determined by a pre-procedure pregnancy test, or women who are breastfeeding
* Class III or IV congestive heart failure
* Myocardial infarction within the last 6 months
* Coronary stenting or cardiac surgery within the last 6 months
* History of unstable angina
* Uncontrolled hypertension
* Intolerance to caffeinated beverages or chocolate
* Dependency on medications that may severely react with caffeine: substrate for Cytochrome P450 1A2 (CYP1A2) (tizanidine), inhibit CYP1A2 (fluvoxamine, ketoconazole, and rofecoxib), induce CYP1A2 (aminoglutethimide, carbamazepine, phenobarbital, and rifampin)
* Enrolment in another study at University of Ottawa Heart Institute (UOHI), unless approved by the Human Ethics Review Board (HREB).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Invasive group: Refractory period of the Right Ventricle (RV) and Right Atrium (RA), Non-Invasive group: Ambulatory monitoring number of atrial and ventricular extrasystoles | Invasive group: Admission to Hospital for the EP study until discharge the same day. Non-Invasive group: From start of 2 consecutive 48 hour ambulatory monitors to their removal.
  Invasive group: During programmed electrical stimulation, determination of the effective refractory period of the atrium and ventricle.
  Non-Invasive group: During Ambulatory Monitoring, determination of atrial and ventricular extrasystoles.

SECONDARY OUTCOMES:
Invasive group: Tachycardia inducibility | Invasive group: Admission to Hospital for the EP study until discharge the same day.
  Invasive group: During programmed electrical stimulation, was SVT induced, was isoproterenol required, and what was the rate of induced tachycardia.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lemery, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Lemery R, Pecarskie A, Bernick J, Williams K, Wells GA. A prospective placebo controlled randomized study of caffeine in patients with supraventricular tachycardia undergoing electrophysiologic testing. J Cardiovasc Electrophysiol. 2015 Jan;26(1):1-6. doi: 10.1111/jce.12504. Epub 2014 Sep 3. PMID 25081280
- Available data/document: Published article — http://onlinelibrary.wiley.com/doi/10.1111/jce.12504/full — DOI: 10.1111/jce.12504